CLINICAL TRIAL: NCT04922580
Title: Predictors of Adverse Neonatal Outcomes in Intrahepatic Cholestasis of Pregnancy
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: maternal and child health hospital of Yong Chuan District (Unknown)
Responsible Party: Principal Investigator, Chen Long,MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: ICP
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalization group: Newborns of ICP mothers require hospitalization after birth
- without Hospitalization group: Newborns of ICP mothers don't require hospitalization after birth

SUMMARY:
Many studies have attempted to find the predictors of adverse neonatal outcome in women with Intrahepatic Cholestasis of Pregnancy(ICP).Serum total bile acid level exceeding 40 µmol/L has been associated with increased risk of meconium staining, low Apgar scores, preterm delivery, and stillbirth.Other predictors such as level of transaminases, history of cholelithiasis, and hepatitis virus infection have been studied but the results are inconclusive.A more comprehensive investigation involving multiple neonatal outcomes and a wide variety of outcome predictors is needed in order to establish guidelines for optimal timing of delivery in pregnancies complicated by ICP. The aim of our study was to evaluate wide variety of predictors of adverse neonatal outcomes in a large cohort of women with ICP .

DETAILED DESCRIPTION:
We performed a retrospective cohort study of all women diagnosed with ICP. Pregnancy outcomes including delivery gestational age, spontaneous preterm delivery, iatrogenic preterm delivery, birth weight, mode of delivery, oligohydramnios, intrauterine growth restriction (IUGR), placental abruption, preterm premature rupture of membrane (PPROM), concerning fetal heart tracing, chorioamnionitis, endometritis, postpartum hemorrhage, transfusion, stillbirth, neonatal intensive care unit (NICU) admission, hyperbilirubinemia, meconium stained amniotic fluid, respiratory distress syndrome(RDS) or transient tachypnea of newborn(TTN) (transient tachypnea of the newborn), and composite neonatal outcome were ascertained. A composite adverse neonatal outcome was created and defined as any of the following: NICU admission, hypoglycemia, hyperbilirubinemia, RDS, TTN, mechanical ventilation use, oxygen by nasal cannula, pneumonia, and stillbirth. PPROM was defined by rupture of membrane before 37 weeks gestation. Concerning fetal heart tracing was defined as recurrent variable or late decelerations with moderate variability, prolonged decelerations, or category 3 tracing. Providers who were caring for the women reviewed and independently characterized fetal heart tracings. Since fetal heart tracings were not accessible to authors, authors accepted the providers' interpretation. For analysis of concerning fetal heart tracing, women with non-labor cesarean section were excluded. Hyperbilirubinemia was defined by neonatal hyperbilirubinemia that required phototherapy. Hypoglycemia was defined by neonatal hypoglycemia that required intravenous infusion. Diagnosis of RDS and TTN were made by the managing neonatologist and based on standard clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Newborns were born in maternal and child health hospital of Yong Chuan District from January 2012 to December 2020;②all Newborns' mothers diagnosed intrahepatic cholestasis of pregnancy.

Exclusion Criteria:

The newborns were born with severe congenital heart disease and deformities

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | up to 28 days
  Hypoglycemia was defined by neonatal hypoglycemia that required intravenous infusion
Hyperbilirubinemia | up to 28 days
  Hyperbilirubinemia was defined by neonatal hyperbilirubinemia that required phototherapy
NICU admission | up to 28 days
  Newborns required hospitalization in the NICU after birth
RDS | up to 28 days
  Newborns were diagnosed with respiratory distress syndrome
TTN | up to 28 days
  Newborns were diagnosed with transient tachypnea of the newborn
mechanical ventilation use | up to 28 days
  Newborns required mechanical ventilation
oxygen by nasal cannula | up to 28 days
  Newborns required oxygen by nasal cannula
pneumonia | up to 28 days
  Newborns were diagnosed with pneumonia
stillbirth | up to 1 day
  newborns died after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided